CLINICAL TRIAL: NCT03338621
Title: An Open-Label, Partially Randomized Trial to Evaluate the Efficacy, Safety and Tolerability of a 4-month Treatment of Bedaquiline Plus Pretomanid Plus Moxifloxacin Plus Pyrazinamide (BPaMZ) Compared to a 6-month Treatment of HRZE/HR (Control) in Adult Participants With Drug-Sensitive Smear-Positive Pulmonary Tuberculosis (DS-TB) and a 6-month Treatment of BPaMZ in Adult Participants With Drug Resistant, Smear-Positive Pulmonary Tuberculosis (DR-TB)
Brief Title: Trial to Evaluate the Efficacy, Safety and Tolerability of BPaMZ in Drug-Sensitive (DS-TB) Adult Patients and Drug-Resistant (DR-TB) Adult Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SimpliciTB (B-Pa-M-Z) NC-008
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis, MDR; Tuberculosis; Drug-Resistant Tuberculosis
Keywords: tuberculosis; drug-resistant tuberculosis; TB; DR-TB; pretomanid; PA-824; bedaquiline; TMC207; moxifloxacin; pyrazinamide; HRZE; TB Alliance; NC-008; drug-sensitive tuberculosis; DS-TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis | interventions — pretomanid; bedaquiline; Moxifloxacin; Pyrazinamide; Isoniazid; Rifampin; Ethambutol

STUDY DESIGN:
Intervention Model Description: Phase 2c multi-center, open-label, partially randomized clinical trial in DS-TB and DR-TB participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Drug Sensitive BPaMZ (Experimental): Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 9 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 17 weeks (Total treatment duration 4 months
  Interventions: Drug: Pretomanid; Drug: Bedaquiline; Drug: Moxifloxacin; Drug: Pyrazinamide
- Drug Sensitive Standard Treatment (Active Comparator): isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg (HRZE) combination tablets for 8 weeks AND isoniazid 75 mg + rifampicin 150 mg (HR) combination tablets for Weeks 9 to 26
  Interventions: Drug: HRZE; Drug: HR
- Drug Resistant BPaMZ (Experimental): Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 18 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 26 weeks (Total treatment duration 6 months)
  Interventions: Drug: Pretomanid; Drug: Bedaquiline; Drug: Moxifloxacin; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Pretomanid — 200 mg tablets
  Other Names: PA-824; Pa
  Arms: Drug Resistant BPaMZ; Drug Sensitive BPaMZ
Drug: Bedaquiline — 100 mg tablets
  Other Names: B; TMC207
  Arms: Drug Resistant BPaMZ; Drug Sensitive BPaMZ
Drug: Moxifloxacin — 400 mg tablets
  Other Names: M
  Arms: Drug Resistant BPaMZ; Drug Sensitive BPaMZ
Drug: Pyrazinamide — 500 mg tablets
  Other Names: Z
  Arms: Drug Resistant BPaMZ; Drug Sensitive BPaMZ
Drug: HRZE — isoniazid 75 mg plus rifampicin 150 mg plus pyrazinamide 400 mg plus ethambutol 275 mg combination tablets
  Other Names: isoniazid; rifampicin; ethambutol
  Arms: Drug Sensitive Standard Treatment
Drug: HR — isoniazid 75 mg plus rifampicin 150 mg combination tablets
  Other Names: isoniazid; rifampicin
  Arms: Drug Sensitive Standard Treatment

SUMMARY:
To evaluate the efficacy, safety and tolerability at 8 weeks (2-months), 52 weeks (12-months), and 104 Weeks (24-months) post the start of the following treatment regimens in participants with: Drug Sensitive TB (DS-TB) patients given BPaMZ for 17 Weeks ( or 4 months) vs. Standard HRZE/HR treatment given for 26 weeks (or 6 months) and Drug Resistant TB (DR-TB) patients given BPaMZ for 26 Weeks (or 6 months)

DETAILED DESCRIPTION:
Phase 2c multi-center, open-label, partially randomized clinical trial in DS-TB and DR-TB participants.

All participants in the below arms will have follow-up for a period of 104 weeks (24 months) from the start of therapy.

Participants with Drug Sensitive TB (DS-TB):

Participants with DS-TB will be randomized to one of two treatment arms. These participants will receive either BPaMZ daily for 17 weeks (4 months), or HRZE/HR combination tablets daily for 26 weeks (6 months). participants will be stratified for co-infection with human immunodeficiency virus (HIV) and cavitation.

Participants with Drug Resistant TB (DR-TB):

Participants with DR-TB will be assigned to receive BPaMZ daily for 26 weeks (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Sputum positive for tubercule bacilli (at least 1+ on the International Union Against Tuberculosis and Lung Disease [IUATLD]/WHO scale (Appendix 1) on smear microscopy) at the trial laboratory.
* Participants with one of the following pulmonary TB conditions:

DS-TB treatment arm participants should be:

* sensitive to rifampicin and isoniazid by rapid sputum based test AND
* either newly diagnosed for TB or have a history of being untreated for at least 3 years after cure from a previous episode of TB.

DR-TB treatment arm participants should be Resistant to rifampicin and/or isoniazid.

* Of non-childbearing potential or willing to practice effective methods of birth control
* Body weight (in light clothing and no shoes) ≥ 30 kg.
* Completed informed consent form

Exclusion Criteria:

* Karnofsky score <60%
* Any risk factor for QT prolongation
* Any planned contraindicated medicines
* Resistant to fluoroquinolones (rapid, sputum-based molecular screening tests).

Any of the following lab toxicities/abnormalities:

* CD4+ count < 100 cells/µL (HIV infected participants)
* platelets <75,000/mm³
* creatinine >1.5 times upper limit of normal (ULN)
* eGFR ≤ 60 mL/min
* haemoglobin <8.0 g/dL
* serum potassium less than the lower limit of normal for the laboratory.
* GGT: greater than 3 x ULN
* AST: ≥3.0 x ULN to be excluded;
* ALT: ≥3.0 x ULN to be excluded
* ALP: ≥3.0 x ULN to be excluded
* Total bilirubin: >1.5 x ULN to be excluded;
* Direct bilirubin: greater than 1x ULN to be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morounfolu Olugbosi, MD MSc, Study Chair — Global Alliance for TB Drug Development
Locations (26):
- Brazil (2):
  - Evandro Chagas, Rio de Janeiro
  - FIOCRUZ, Rio de Janeiro
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Institut Perubatan Respiratori, Kuala Lumpur, Malaysia
- Philippines (2):
  - Lung Center of Philippines, Manila
  - Tropical Disease Foundation, Manila
- Russia (5):
  - Moscow City Research and Practice Tuberculosis Treatment Centre, Moscow
  - Central TB Research Institute of the Federal Agency of Scientific Organizations, Moscow
  - Research Institute of Phthisiopulmonology of I. M. Sechenov First Moscow State Medical University, Moscow
  - Research Institute of the Phthisiopulmonology, Saint Petersburg
  - Ural Research Institute of Phthisiopulmonology, Yekaterinburg
- South Africa (10):
  - THINK, Pietermaritzburg, KwaZulu-Natal
  - Madibeng Centre for Research, Brits
  - TASK, Cape Town
  - University of Cape Town Lung Institute, Cape Town
  - Enhancing Care Foundation, Durban
  - CHRU, King Dinuzulu, Durban
  - CHRU, Helen Joseph Hospital, Johannesburg
  - PHRU, Tshepong Hospital, Klerksdorp
  - CHRU, Empilweni TB Hospital, Port Elizabeth
  - Setshaba Research Centre, Soshanguve
- Tanzania (4):
  - Ifakara Health Institute, Bagamoyo
  - NIMR-Mbeya, Mbeya
  - Kilimanjaro Clinical Research Institute, Moshi
  - Mwanza Intervention Trials Unit, Mwanza
- Case Western Reserve University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
IPD from the trial will be submitted to Critical Path Institute which will make fully anonymized data available through the Tuberculosis Platform for Aggregation of Clinical TB Studies (TB-PACTS) database. Data sets for Drug susceptibility data, Demographic data, MTB diagnostic testing results, Concomitant medications information, Adverse event information, Treatment adherence information, Co-morbidities, Treatment outcomes, HIV co-infection information, CD4 counts, TB disease symptoms from all collected IPD will be made available.
Time Frame: Data is expected to become available in mid-2024.
Access Criteria: Researchers must agree to the Terms and Conditions for Use of the TB-PACTS data platform and submit an online application form to request access to the data platform.
URL: https://c-path.org/tools-platforms/tb-pacts/

REFERENCES:
- [Derived] Cevik M, Thompson LC, Upton C, Rolla VC, Malahleha M, Mmbaga B, Ngubane N, Abu Bakar Z, Rassool M, Variava E, Dawson R, Staples S, Lalloo U, Louw C, Conradie F, Eristavi M, Samoilova A, Skornyakov SN, Ntinginya NE, Haraka F, Praygod G, Mayanja-Kizza H, Caoili J, Balanag V, Dalcolmo MP, McHugh T, Hunt R, Solanki P, Bateson A, Crook AM, Fabiane S, Timm J, Sun E, Spigelman M, Sloan DJ, Gillespie SH; SimpliciTB Consortium. Bedaquiline-pretomanid-moxifloxacin-pyrazinamide for drug-sensitive and drug-resistant pulmonary tuberculosis treatment: a phase 2c, open-label, multicentre, partially randomised controlled trial. Lancet Infect Dis. 2024 Sep;24(9):1003-1014. doi: 10.1016/S1473-3099(24)00223-8. Epub 2024 May 17. PMID 38768617

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug Sensitive-TB 4BPaMZ: Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 9 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 17 weeks (Total treatment duration 4 months)
  Pretomanid: 200 mg tablets
  Bedaquiline: 100 mg tablets
  Moxifloxacin: 400 mg tablets
  Pyrazinamide: 500 mg tablets
- Drug Sensitive-TB 2HRZE/4HR: isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg (HRZE) combination tablets for 8 weeks AND isoniazid 75 mg + rifampicin 150 mg (HR) combination tablets for Weeks 9 to 26
  HRZE: isoniazid 75 mg plus rifampicin 150 mg plus pyrazinamide 400 mg plus ethambutol 275 mg combination tablets
  HR: isoniazid 75 mg plus rifampicin 150 mg combination tablets
  Participant Dosage based on weight
- Drug Resistant-TB 6BPaMZ: Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 18 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 26 weeks (Total treatment duration 6 months)
  Pretomanid: 200 mg tablets
  Bedaquiline: 100 mg tablets
  Moxifloxacin: 400 mg tablets
  Pyrazinamide: 500 mg tablets
Period: Overall Study
Arm/Group | Drug Sensitive-TB 4BPaMZ | Drug Sensitive-TB 2HRZE/4HR | Drug Resistant-TB 6BPaMZ
Started | 150 | 153 | 152
Completed | 121 | 134 | 117
Not Completed | 29 | 19 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Sensitive-TB 4BPaMZ | Drug Sensitive-TB 2HRZE/4HR | Drug Resistant-TB 6BPaMZ | Total
Number analyzed (Participants) | 150 | 153 | 152 | 455
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 36.4 [25.0 to 45.0] | 36.3 [26.0 to 46.0] | 37.6 [26.0 to 47.0] | 36.7 [26.0 to 46.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 58 | 131
  Male | 112 | 118 | 94 | 324
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 3 | 13 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 108 | 119 | 82 | 309
  White | 29 | 25 | 31 | 85
  More than one race | 5 | 6 | 26 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 6 | 2 | 9 | 17
  Tanzania | 52 | 48 | 7 | 107
  Brazil | 4 | 3 | 28 | 35
  South Africa | 56 | 68 | 72 | 196
  Uganda | 3 | 6 | 8 | 17
  Malaysia | 2 | 1 | 4 | 7
  Georgia | 23 | 20 | 9 | 52
  Russia | 4 | 5 | 15 | 24
Height [Mean (Inter-Quartile Range); unit: cm] | 168.1 [163.0 to 175.0] | 168.9 [163.0 to 175.0] | 167.8 [162.0 to 175.0] | 168.3 [162.0 to 175.0]
Weight [Mean (Inter-Quartile Range); unit: kg] | 56.5 [48.8 to 62] | 55.6 [49.0 to 59.0] | 56.6 [48.3 to 63.6] | 56.3 [48.5 to 61.5]
BMI [Mean (Inter-Quartile Range); unit: Kg/m^2] | 20.0 [17.6 to 21.4] | 19.5 [17.2 to 20.4] | 20.1 [17.1 to 22.2] | 19.9 [17.3 to 21.2]
HIV Status [Count of Participants; unit: Participants]
  Positive | 25 | 27 | 35 | 87
  Negative | 125 | 126 | 117 | 368
Smoking [Count of Participants; unit: Participants]
  Never | 59 | 49 | 72 | 180
  Current | 59 | 64 | 39 | 162
  Former | 32 | 40 | 41 | 113
Alcohol Use [Count of Participants; unit: Participants]
  Never | 37 | 42 | 55 | 134
  Current | 63 | 69 | 48 | 180
  Former | 50 | 42 | 49 | 141
Previous Tuberculosis (TB) diagnoses [Number; unit: participants] — One participant can select more than one type of TB for disease history. Extensively drug-resistant TB (XDR-TB) was based on the pre-2021 WHO definition
  participants
    Drug Sensitive (DS-TB) | 150 | 153 | 33 | 336
    Mono-resistant TB | 0 | 0 | 45 | 45
    Multi-drug Resistant (MDR-TB) | 0 | 0 | 99 | 99
    Pre-extensively Resistant (Pre-XDR TB) | 0 | 0 | 1 | 1
    Extensively Resistant (XDR-TB) | 0 | 0 | 2 | 2
Screening smear microscopy for Acid Fast Bacilli (AFB) [Count of Participants; unit: Participants]
  No AFB seen | 0 | 0 | 0 | 0
  Scanty Positive | 0 | 0 | 0 | 0
  1+ | 20 | 28 | 37 | 85
  2+ | 49 | 53 | 47 | 149
  3+ | 81 | 72 | 67 | 220
  Missing | 0 | 0 | 1 | 1
Time to positive at baseline [Mean (Inter-Quartile Range); unit: days] | 5.4 [3.9 to 6.2] | 5.8 [4.2 to 6.5] | 7.4 [4.7 to 8.9] | 6.2 [4.2 to 7.2]
Chest x-ray at Screening [Count of Participants; unit: Participants]
  Normal | 5 | 2 | 7 | 14
  Abnormal | 145 | 151 | 144 | 440
  Missing | 0 | 0 | 1 | 1
Chest X-Ray Cavities at Screening [Count of Participants; unit: Participants]
  None | 31 | 37 | 31 | 99
  Unilateral | 75 | 76 | 70 | 221
  Bilateral | 44 | 40 | 50 | 134
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Culture Negative Status by 8 Weeks
Description: Culture negative status is achieved when a participant produces at least two negative culture results at different visits (at least 7 days apart) without an intervening positive culture result for M.tb.
Time Frame: Days 0-56 (8 weeks)
Population: Limited to Drug Sensitive TB groups. Participants were considered unassessable and therefore excluded from the Modified Intent to Treat (MITT) population if they were late exclusion or if they did not have culture confirmation of M.tb at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Sensitive-TB 2HRZE/4HR | Drug Sensitive-TB 4BPaMZ
Number analyzed (Participants) | 148 | 145
Participants | 70 | 122
Statistical Analysis 1: Comparison: Drug Sensitive-TB 2HRZE/4HR vs Drug Sensitive-TB 4BPaMZ; Test type: Superiority; p < 0.001, Log Rank; Cox Proportional Hazard = 2.93, 95% CI 2-sided [2.17 to 3.96]

2. Secondary Outcome: Number of Participants With Bacteriologic Failure or Relapse or Clinical Failure (Unfavorables) at 52 Weeks From Start of Therapy (12 Months)
Description: Unfavorable status:
  1. Participants not classified as having achieved or maintained culture negative status when last seen
  2. Participants previously classified as having culture negative status who, following the end of treatment, have two positive cultures without an intervening negative culture
  3. Participants who had a positive culture not followed by at least two negative cultures when last seen
  4. Participants dying from any cause during treatment, except from violent or accidental cause, not including suicide
  5. Participants definitely or possibly dying from TB related cause during the follow-up phase
  6. Participants requiring an extension of their treatment beyond that permitted by the protocol a restart or a change of treatment for any reason except reinfection or pregnancy
  7. Participants lost to follow up or withdrawn from the study before end of treatment
Time Frame: 52 weeks after start of therapy
Population: TB Specific Modified Intent to Treat (TB-MITT) population participants were unassessable and excluded if they were a late exclusion, became pregnant and stopped treatment, had suspected or confirmed COVID-19 and stopped treatment, died during treatment from violent or accidental cause, died during follow-up with no evidence of TB, reinfected with a different strain of TB, had contaminated or missing sputum samples at the endpoint visit (and able to produce sputum).
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Sensitive-TB 4BPaMZ | Drug Sensitive-TB 2HRZE/4HR | Drug Resistant-TB 6BPaMZ
Number analyzed (Participants) | 144 | 144 | 133
Participants
  Favorable | 120 | 134 | 111
  Unfavorable | 24 | 10 | 22

3. Secondary Outcome: Time to Culture Negative Status
Description: Culture conversion is a diagnostic criteria indicating the point at which samples taken from a patient infected with a tuberculosis can no longer produce tuberculosis cell cultures, that point is considered culture negativity
Time Frame: During treatment (17 or 26 weeks)
Population: Participants were unassessable and excluded from the Modified Intent to Treat (MITT) population if they were a late exclusions.
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Drug Sensitive-TB BPaMZ: Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 9 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 17 weeks (Total treatment duration 4 months
  Pretomanid: 200 mg tablets
  Bedaquiline: 100 mg tablets
  Moxifloxacin: 400 mg tablets
  Pyrazinamide: 500 mg tablets
- Drug Sensitive-TB 2HRZE/4HR: isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg (HRZE) combination tablets for 8 weeks AND isoniazid 75 mg + rifampicin 150 mg (HR) combination tablets for Weeks 9 to 26
  HRZE: isoniazid 75 mg plus rifampicin 150 mg plus pyrazinamide 400 mg plus ethambutol 275 mg combination tablets
  HR: isoniazid 75 mg plus rifampicin 150 mg combination tablets
- Drug Resistant-TB BPaMZ: Bedaquiline 200 mg daily for 8 weeks then 100 mg daily for 18 weeks, together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg daily for 26 weeks (Total treatment duration 6 months)
  Pretomanid: 200 mg tablets
  Bedaquiline: 100 mg tablets
  Moxifloxacin: 400 mg tablets
  Pyrazinamide: 500 mg tablets
Arm/Group | Drug Sensitive-TB BPaMZ | Drug Sensitive-TB 2HRZE/4HR | Drug Resistant-TB BPaMZ
Number analyzed (Participants) | 145 | 148 | 133
weeks | 6 [4 to 8] | 11 [6 to 12] | 5 [3 to 7]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: All listed adverse events (AEs) are treatment emergent adverse events (TEAE) which are defined as AEs that started or worsened at or after the first administration of study drug up to and including 14 days after the last study drug administration.
Arm/Group | Drug Sensitive-TB BPaMZ | Drug Sensitive-TB 2HRZE/4HR | Drug Resistant-TB BPaMZ
All-Cause Mortality (participants affected / at risk) | 3/150 | 2/153 | 4/149
Serious Adverse Events (participants affected / at risk) | 17/150 | 7/153 | 16/149
Other Adverse Events (participants affected / at risk) | 139/150 | 144/153 | 142/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Sensitive-TB BPaMZ (N=150) | Drug Sensitive-TB 2HRZE/4HR (N=153) | Drug Resistant-TB BPaMZ (N=149)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Cor Pulmonae (Cardiac disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 8 | 1 | 4
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Psoas Abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 2 | 0
Electrocardiogram ST Segment Elevation (Investigations) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 2 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Post-Traumatic Epilepsy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Plueral Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Physical Assault (Social circumstances) | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Sensitive-TB BPaMZ (N=150) | Drug Sensitive-TB 2HRZE/4HR (N=153) | Drug Resistant-TB BPaMZ (N=149)
Anemia (Blood and lymphatic system disorders) | 9 | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 5 | 18
Gastritis (Gastrointestinal disorders) | 12 | 0 | 12
Nausea (Gastrointestinal disorders) | 21 | 5 | 22
Vomiting (Gastrointestinal disorders) | 11 | 7 | 18
Pyrexia (General disorders) | 9 | 4 | 3
Hepatotoxicity (Hepatobiliary disorders) | 10 | 3 | 7
Conjunctivitis (Infections and infestations) | 3 | 0 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 12 | 10
Urinary Tract Infection (Infections and infestations) | 10 | 14 | 5
Alanine Aminotransferase Increased (Investigations) | 14 | 10 | 8
Aspartate Aminotransferase Increased (Investigations) | 10 | 9 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 5 | 11 | 0
Hepatic Enzyme Increased (Investigations) | 18 | 14 | 11
Lipase Increased (Investigations) | 6 | 8 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 2 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 8 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 23 | 25 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 73 | 69 | 43
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 24 | 34
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 9 | 3
Dizziness (Nervous system disorders) | 7 | 4 | 18
Headache (Nervous system disorders) | 10 | 14 | 18
Neuropathy Peripheral (Nervous system disorders) | 5 | 11 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish, present or use the Study Data for its own instruction, research or publication without the prior express written consent of Sponsor. Because the Study is funded, in whole or in part, by the Bill and Melinda Gates Foundation (the "Foundation"), all peer-reviewed published research relating to the Study must comply with the Foundation's Open Access Policy.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT03338621/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03338621/SAP_001.pdf